CLINICAL TRIAL: NCT05584345
Title: EFFECTS OF BREATHING EXERCISES ON PAIN AND FUNCTIONALITY IN ROTATOR CUFF TEARS: A RANDOMIZED CONTROLLED TRIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-240
Record Dates: First submitted 2022-09-20; First posted 2022-10-18 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Syndrome
Keywords: respiratory exercises; rotator cuff syndrome; pain
MeSH Terms: conditions — Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy (Active Comparator): Traditional physiotherapy applications will be applied.
  Interventions: Other: Conventional Treatment and manual therapy
- breathing exercises and conventional therapy program (Experimental): In addition to traditional physiotherapy, respiratory exercises will be applied.
  Interventions: Other: Manual therapy and Respiratory Exercises

INTERVENTIONS:
Other: Conventional Treatment and manual therapy — Cold pack, ultrasound, TENS, finger ladder, Codman, shoulder wheel, and Wand exercises, as well as stretching and capsule exercises, will be used in addition to conventional physiotherapy. There will be 30 repetitions in each direction of the Codman exercises. 5 days a week, for a total of 30 sessions, the afflicted shoulder will get 6 minutes of daily US treatment, with complete contact to the shoulder area and at a right angle. All patients will receive manual stretching in the shoulder flexion, abduction, extension, external rotation, and internal rotation directions. In addition, participants will receive manual therapy techniques, including Glenohumeral joint (GH) distraction, glenohumeral joint inferior gliding, anterior gliding, and posterior gliding, scapulothoracic joint distraction, scapulothoracic joint superior, inferior, medial, and lateral gliding. Each manual therapy technique was performed with 10 repetitions per participant
  Arms: Conventional therapy
Other: Manual therapy and Respiratory Exercises — In addition to the treatment program applied in conventional therapy and manual therapy,, participants in this group also will perform diaphragmatic breathing exercises, pursed-lip breathing exercises, and relaxation breathing exercises. Each breathing exercise will be performed with 10 repetitions under physiotherapist supervision. Participants were also asked to continue the breathing exercises at home, performing them three times a day with 10 repetitions per session for a duration of six weeks.
  Arms: breathing exercises and conventional therapy program

SUMMARY:
As it causes pain and disability in individuals with rotator cuff lesions, which is one of the most common causes of shoulder pain, it affects performance in activities of daily living. Shoulder pain significantly affects the quality of life of individuals. The aim of conventional treatment in Rotator Cuff injuries is to reduce the inflammation in the area and to enable the shoulder to perform its normal functions. Conventional treatment is to restore muscle balance in the shoulder area. Muscle balance is achieved by strengthening the teres minor, infraspinatus, and subscapularis, which are also the humeral head depressors, and by strengthening the serratus anterior, levator scapula. For strengthening, the shoulder must have a full range of motion. In our study, stretching exercises, cold pack, Ultrasound, TENS, wand, and Codman exercises, which are classical physiotherapy methods, will be applied to all three groups. There are also studies in the literature investigating the effects of traditional physiotherapy methods on individuals with shoulder Rotator Cuff syndrome. The benefits of breathing exercises on pain, shoulder joint range of motion, and balance have all been researched in the literature. Increased diaphragm activity also guarantees that posture and body positions are maintained healthily. Diaphragm activity generally alters how an individual perceives pain. Diaphragmatic breathing is a therapeutic approach for musculoskeletal disorders.

DETAILED DESCRIPTION:
Breathing techniques have been demonstrated to reduce shoulder pain and increase ROM at the literature. However, no study has been found on the effectiveness of breathing exercises applied in addition to conventional physiotherapy in individuals with Rotator Cuff syndrome.

Based on all of this knowledge, it was designed for this study to examine the efficacy of breathing exercises used in combination with traditional physiotherapy in patients with Rotator Cuff syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. The participants were between the ages of 30 and 55
2. No history of shoulder surgery
3. Exhibited restricted shoulder joint range of motion,
4. A diagnosed rotator cuff tear

Exclusion Criteria:

1. individuals with a history of significant shoulder trauma
2. anatomical deformities, skeletal fractures, diagnosed orthopedic or rheumatologic disorders, participation in a physiotherapy program within the last six months
3. Presence of a cardiac pacemaker, current infections, recent myocardial infarction (within the last six months), or any other condition that could interfere with their ability to perform the prescribed exercises

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Visual Analog scale (VAS) | From enrollment to the end of treatment at six weeks
  Pain intensity will be with VAS that is a tool commonly used to assess the intensity of musculoskeletal pain (18). The VAS will be used to evaluate the level of shoulder pain experienced by participants at rest, and during activity. Participants were asked to rate their pain intensity on a scale ranging from 0 to 10, where 0 indicates "no pain" and 10 indicates "worst possible pain." The participants' responses will be recorded in the case report forms.

SECONDARY OUTCOMES:
Goniometric Measurement | From enrollment to the end of treatment at six weeks
  In our study, the degrees of flexion, extension, abduction, internal rotation, and external rotation of the affected shoulder will be measured by means of a universal goniometer. Flexion and abduction 0-180 degrees, extension 45 degrees, internal and external rotation 0-90 degrees will be taken as reference.
DASH | From enrollment to the end of treatment at six weeks
  The DASH scale, created by the American Academy of Orthopedic Surgeons in collaboration with other professional organizations, is a standardized instrument used to evaluate physical limitations and functional impairments in individuals with upper extremity conditions. The DASH questionnaire includes three distinct subdomains. The first section consists of 30 questions, with 21 items focusing on the patient's difficulties in performing daily activities, five items assessing symptoms, and the remaining four items addressing social functioning, work productivity, sleep quality, and self-confidence. Higher scores on the DASH questionnaire indicate greater levels of disability and functional limitation, whereas lower scores reflect less disability and better functional status

CONTACTS AND LOCATIONS:
Overall Officials: BURAK MENEK, PhD, Principal Investigator — Medipol University; UMUT İSLAM TAYBOĞA, RA, Principal Investigator — Medipol University; Sule Ayan, Msc, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)